CLINICAL TRIAL: NCT03358654
Title: Evaluating the Safety and Efficacy of Mesenchymal Stem Cells From Umbilical Cord in the Treatment of Knee Joint Osteoarthritis
Brief Title: Evaluating Safety and Efficacy of Mesenchymal Stem Cells From Umbilical Cord
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, yangziyi, arthritis clinic and research center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUPH20170911
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Umbilical Cord Bleeding; Knee Osteoarthritis
Keywords: Umbilical Cord Bleeding; Knee Osteoarthritis; stem cells
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesenchymal stem cells (Experimental): Inject mesenchymal stem cells from umbilical cord. The patients will be followed up at 1, 2, 3, and 6 months after the injection
  Interventions: Drug: mesenchymal stem cells from umbilical cord

INTERVENTIONS:
Drug: mesenchymal stem cells from umbilical cord — inject mesenchymal stem cells from umbilical cord，and the patients will be followed up at 1, 2, 3, and 6 months after the injection.

SUMMARY:
This study was to evaluate the safety and efficacy of Mesenchymal Stem Cells (MSCs) from umbilical cord in the treatment of 7 knee OA patients by assessing unexplained local and systemic symptoms or death before and at 1, 2, 3, 6 months after the injection.

DETAILED DESCRIPTION:
This is a single group assignment study with a total of 9 knee osteoarthritis patients participants. All of the patients will receive the anticular injection with MSCs from umbilical cord and unexplained local and systemic symptoms or death before the end of following-up will be assessed to evaluate the safety and efficacy of mesenchymal stem cells from umbilical cord.

ELIGIBILITY:
Inclusion Criteria:

① K / L score of 2-3; ② chronic knee pain; ③ no local or systemic infection; ④ without obvious contraindication of the joint puncture from hematology and biochemical tests; ⑤ informed consent. -

Exclusion Criteria:

① older than 75 years old or less than 18 years old, or without full capacity for civil conduct; ② HIV, hepatitis virus or syphilis virus infection or their serology is positive; ③ BMI index is greater than 30; ④ congenital or acquired knee deformity; ⑤ pregnant or lactating women; ⑥ tumor patients; ⑦ immunodeficiency patients; ⑧ intra-articular drug injection history within 3 months; ⑨ participating in other clinical trials; ⑩ other patients who researchers believe are not eligible for inclusion such as suffering from other concomitant diseases. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Unexplained local and systemic symptoms or death | 6 months
  The severity of AE must be recorded and graded according to the CTCAE criteria, and its relationship to therapy must be assessed according to the following definition:①not related: there is evidence that the cause of adverse events is not due to intra-articular injection therapy (such as previous conditions, potential diseases, concurrent diseases); ②related: AE and intra-articular injection are time-related and it is known or suspected that intra-articular injection of drugs can cause the AE; ③it can't be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritis clinic and research center